CLINICAL TRIAL: NCT02443740
Title: A Phase 1, Randomized, Double Blind, Placebo Controlled Study To Investigate The Safety, Tolerability, Pharmacokinetics And Relative Bioavailability Of Single Escalating Oral Doses Of Pf-05251749 In Healthy Adult Subjects
Brief Title: Safety, Tolerability and Pharmacokinetics of BIIB118 (PF-05251749)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: B8001001; SAD (Other: Alias Study Number)
Record Dates: First submitted 2015-05-01; First posted 2015-05-14 (Estimated); Results first posted 2018-05-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Healthy
Keywords: First in human; Single Ascending Dose Study; Safety and Tolerability; Pharmacokinetics; Plasma; Cerebrospinal Fluid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Single Ascending Dose-1 (Part A) (Experimental): Single ascending doses of BIIB118 administered to healthy volunteers in a cross over study design
  Interventions: Drug: BIIB118
- Single Ascending Dose-2 (Part A) (Experimental): Single ascending doses of BIIB118 administered to healthy volunteers in a cross over study design
  Interventions: Drug: BIIB118
- Single Dose Cerebrospinal Fluid (Part B) (Experimental): Single maximum dose from Part A of BIIB118 administered to healthy volunteers to assess the PK of BIIB118 in CSF
  Interventions: Drug: BIIB118

INTERVENTIONS:
Drug: BIIB118 — Single ascending doses of BIIB118 as extemporaneously prepared solution/suspension, once every 2 week in a cross over study: 3 mg, 30 mg, 200 mg, 800 mg and placebo
  Other Names: PF-05251749
  Arms: Single Ascending Dose-1 (Part A)
Drug: BIIB118 — Single ascending doses of BIIB118 as extemporaneously prepared solution/suspension, once every 2 week in a cross over study: 10 mg, 100 mg, 400 mg, and placebo
  Other Names: PF-05251749
  Arms: Single Ascending Dose-2 (Part A)
Drug: BIIB118 — Single dose (Maximum Tolerated Dose) of BIIB118 as extemporaneously prepared solution/suspension
  Other Names: PF-05251749
  Arms: Single Dose Cerebrospinal Fluid (Part B)

SUMMARY:
This is a First in human (FIH) single ascending dose study to evaluate the safety, tolerability and pharmacokinetics (PKs) of BIIB118 following single oral doses in healthy human subjects

DETAILED DESCRIPTION:
This study was previously posted by Pfizer. In March, 2020, sponsorship of the trial was transferred to Biogen.

ELIGIBILITY:
Inclusion Criteria:

•Healthy male and/or female subjects of non-childbearing potential between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests).

Female subjects of non-childbearing potential must meet at least one of the following criteria:

1. Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; and have a serum follicle-stimulating hormone (FSH) level confirming the post-menopausal state;
2. Have undergone a documented hysterectomy and/or bilateral oophorectomy;
3. Have medically confirmed ovarian failure. All other female subjects (including females with tubal ligations and females that do NOT have a documented hysterectomy, bilateral oophorectomy and/or ovarian failure) will be considered to be of childbearing potential.

   * Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
   * Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
   * Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study medication (whichever is longer).
* Screening supine blood pressure >= 140 mm Hg (systolic) or >=90 mm Hg (diastolic), following at least 5 minutes of rest. If BP is >=140 mm Hg (systolic) or >=90 mm Hg (diastolic), repeat per local standard operating procedures (SOP). If orthostatic changes are present and deemed to be clinically significant by the investigator, Subject can be excluded.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2015-05-31 (Actual); Primary Completion 2015-10-31 (Actual); Study Completion 2015-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B8001001&StudyName=A%20Phase%201%2C%20Randomized%2C%20Double%20Blind%2C%20Placebo%20Controlled%20Study%20To%20Investigate%20The%20Safety%2C%20Tolerability%2C%20Pharmacokinetics%20And%20Relative%20Bioavailability%20Of%20Single%20Escalating%20Oral%20Doses%20Of%20Pf-05251749%20In%20Healthy%20Adult%20Subjects

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of 4 cohorts. Cohort 1 and 2 was a 4 period crossover sequence of PF-05251749 and matching placebo. Cohort 3 was designed to characterize the pharmacokinetic (PK) of PF-05251749 in cerebrospinal fluid (CSF) samples. Cohort 4 was a 2 period crossover sequence of unmilled and milled PF-05251749.
Groups:
- Cohort 1 PF-05251749: Placebo + 30 mg + 250 mg + 500 mg: Participants received a single oral dose of PF-05251749 suspension on Day 1 of each Intervention Period (4 Intervention Periods of 3 days each). Participants received study treatment in following sequences: Placebo, PF-05251749 30 milligram (mg), 250 mg and 500 mg in Intervention Period 1, 2, 3 and 4 respectively. All doses were administered in fasted state except PF-05251749 500 mg. A washout period of at least 7 days was maintained between each Intervention Period.
- Cohort 1 PF-05251749: 3 mg + Placebo + 250 mg + 500 mg: Participants received a single oral dose of PF-05251749 suspension on Day 1 of each Intervention Period (4 Intervention Periods of 3 days each). Participants received study treatment in following sequences: PF-05251749 3 mg, placebo, PF-05251749 250 mg and 500 mg in Intervention Period 1, 2, 3 and 4 respectively. All doses were administered in fasted state except PF-05251749 500 mg. A washout period of at least 7 days was maintained between each Intervention Period.
- Cohort 1 PF-05251749: 3 mg + 30 mg + Placebo + 500 mg: Participants received a single oral dose of PF-05251749 suspension on Day 1 of each Intervention Period (4 Intervention Periods of 3 days each). Participants received study treatment in following sequences: PF-05251749 3 mg, 30 mg, placebo and PF-05251749 500 mg in Intervention Period 1, 2, 3 and 4 respectively. All doses were administered in fasted state except PF-05251749 500 mg. A washout period of at least 7 days was maintained between each Intervention Period.
- Cohort 1 PF-05251749: 3 mg + 30 mg + 250 mg + Placebo: Participants received a single oral dose of PF-05251749 suspension on Day 1 of each Intervention Period (4 Intervention Periods of 3 days each). Participants received study treatment in following sequences: PF-05251749 3 mg, 30 mg, 250 mg and placebo in Intervention Period 1, 2, 3 and 4 respectively. All doses were administered in fasted state except PF-05251749 500 mg. A washout period of at least 7 days was maintained between each Intervention Period.
- Cohort 2 PF-05251749: Placebo + 100 mg + 500 mg + 1000 mg: Participants received a single oral dose of PF-05251749 suspension on Day 1 of each Intervention Period (4 Intervention Periods of 3 days each). Participants received study treatment in following sequences: PF-05251749 placebo, PF-05251749 100 mg, PF-05251749 500 mg, PF-05251749 1000 mg in Intervention Period 1, 2, 3 and 4 respectively. All doses were administered in fasted state. A washout period of at least 7 days was maintained between each Intervention Period.
- Cohort 2 PF-05251749: 10 mg + Placebo + 500 mg + 1000 mg: Participants received a single oral dose of PF-05251749 suspension on Day 1 of each Intervention Period (4 Intervention Periods of 3 days each). Participants received study treatment in following sequences: PF-05251749 10 mg, PF-05251749 placebo, PF-05251749 500 mg, PF-05251749 1000 mg in Intervention Period 1, 2, 3 and 4 respectively. All doses were administered in fasted state. A washout period of at least 7 days was maintained between each Intervention Period.
- Cohort 2 PF-05251749: 10 mg + 100 mg + Placebo + 1000 mg: Participants received a single oral dose of PF-05251749 suspension on Day 1 of each Intervention Period (4 Intervention Periods of 3 days each). Participants received study treatment in following sequences: PF-05251749 10 mg, PF-05251749 100 mg, PF-05251749 placebo, PF-05251749 1000 mg in Intervention Period 1, 2, 3 and 4 respectively. All doses were administered in fasted state. A washout period of at least 7 days was maintained between each Intervention Period.
- Cohort 2 PF-05251749: 10 mg + 100 mg + 500 mg + Placebo: Participants received a single oral dose of PF-05251749 suspension on Day 1 of each Intervention Period (4 Intervention Periods of 3 days each). Participants received study treatment in following sequences: PF-05251749 10 mg, PF-05251749 100 mg, PF-05251749 500 mg, PF-05251749 placebo in Intervention Period 1, 2, 3 and 4 respectively. All doses were administered in fasted state. A washout period of at least 7 days was maintained between each Intervention Period.
- Cohort 3 PF-05251749: 500 mg: Participants received a single oral dose of PF-05251749 500 mg suspension on Day 1. CSF samples were collected for a total of 10 hours beginning 2 hours predose and 8 hours post dose.
- Cohort 4 PF-05251749: 500 mg Unmilled + 500 mg Milled: Participants received a single oral dose of PF-05251749 suspension on Day 1 of each Intervention Period (2 Intervention Periods of 3 days each). Participants received study treatment in following sequences: PF-05251749 500mg unmilled, PF-05251749 500mg milled in Intervention Period 1 and 2. All doses were administered in fasted state. A washout period of at least 7 days was maintained between each Intervention Period.
- Cohort 4 PF-05251749: 500 mg Milled + 500 mg Unmilled: Participants received a single oral dose of PF-05251749 suspension on Day 1 of each Intervention Period (2 Intervention Periods of 3 days each). Participants received study treatment in following sequences: PF-05251749 500 mg milled, PF-05251749 500 mg unmilled in Intervention Period 1 and 2. All doses were administered in fasted state. A washout period of at least 7 days was maintained between each Intervention Period.
Period: Intervention Period 1 (3 Days)
Arm/Group | Cohort 1 PF-05251749: Placebo + 30 mg + 250 mg + 500 mg | Cohort 1 PF-05251749: 3 mg + Placebo + 250 mg + 500 mg | Cohort 1 PF-05251749: 3 mg + 30 mg + Placebo + 500 mg | Cohort 1 PF-05251749: 3 mg + 30 mg + 250 mg + Placebo | Cohort 2 PF-05251749: Placebo + 100 mg + 500 mg + 1000 mg | Cohort 2 PF-05251749: 10 mg + Placebo + 500 mg + 1000 mg | Cohort 2 PF-05251749: 10 mg + 100 mg + Placebo + 1000 mg | Cohort 2 PF-05251749: 10 mg + 100 mg + 500 mg + Placebo | Cohort 3 PF-05251749: 500 mg | Cohort 4 PF-05251749: 500 mg Unmilled + 500 mg Milled | Cohort 4 PF-05251749: 500 mg Milled + 500 mg Unmilled
Started | 2 | 2 | 2 | 3 | 2 | 4 | 3 | 2 | 6 | 3 | 3
Completed | 1 | 2 | 2 | 3 | 2 | 2 | 2 | 2 | 6 | 3 | 3
Not Completed | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 1 (7 Days)
Arm/Group | Cohort 1 PF-05251749: Placebo + 30 mg + 250 mg + 500 mg | Cohort 1 PF-05251749: 3 mg + Placebo + 250 mg + 500 mg | Cohort 1 PF-05251749: 3 mg + 30 mg + Placebo + 500 mg | Cohort 1 PF-05251749: 3 mg + 30 mg + 250 mg + Placebo | Cohort 2 PF-05251749: Placebo + 100 mg + 500 mg + 1000 mg | Cohort 2 PF-05251749: 10 mg + Placebo + 500 mg + 1000 mg | Cohort 2 PF-05251749: 10 mg + 100 mg + Placebo + 1000 mg | Cohort 2 PF-05251749: 10 mg + 100 mg + 500 mg + Placebo | Cohort 3 PF-05251749: 500 mg | Cohort 4 PF-05251749: 500 mg Unmilled + 500 mg Milled | Cohort 4 PF-05251749: 500 mg Milled + 500 mg Unmilled
Started | 1 | 2 | 2 | 3 | 2 | 2 | 2 | 2 | 0 | 3 | 3
Completed | 1 | 2 | 2 | 3 | 2 | 2 | 2 | 2 | 0 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Intervention Period 2 (3 Days)
Arm/Group | Cohort 1 PF-05251749: Placebo + 30 mg + 250 mg + 500 mg | Cohort 1 PF-05251749: 3 mg + Placebo + 250 mg + 500 mg | Cohort 1 PF-05251749: 3 mg + 30 mg + Placebo + 500 mg | Cohort 1 PF-05251749: 3 mg + 30 mg + 250 mg + Placebo | Cohort 2 PF-05251749: Placebo + 100 mg + 500 mg + 1000 mg | Cohort 2 PF-05251749: 10 mg + Placebo + 500 mg + 1000 mg | Cohort 2 PF-05251749: 10 mg + 100 mg + Placebo + 1000 mg | Cohort 2 PF-05251749: 10 mg + 100 mg + 500 mg + Placebo | Cohort 3 PF-05251749: 500 mg | Cohort 4 PF-05251749: 500 mg Unmilled + 500 mg Milled | Cohort 4 PF-05251749: 500 mg Milled + 500 mg Unmilled
Started | 1 | 2 | 2 | 3 | 2 | 2 | 2 | 2 | 0 | 3 | 3
Completed | 1 | 2 | 2 | 3 | 2 | 2 | 2 | 2 | 0 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 2 (7 Days)
Arm/Group | Cohort 1 PF-05251749: Placebo + 30 mg + 250 mg + 500 mg | Cohort 1 PF-05251749: 3 mg + Placebo + 250 mg + 500 mg | Cohort 1 PF-05251749: 3 mg + 30 mg + Placebo + 500 mg | Cohort 1 PF-05251749: 3 mg + 30 mg + 250 mg + Placebo | Cohort 2 PF-05251749: Placebo + 100 mg + 500 mg + 1000 mg | Cohort 2 PF-05251749: 10 mg + Placebo + 500 mg + 1000 mg | Cohort 2 PF-05251749: 10 mg + 100 mg + Placebo + 1000 mg | Cohort 2 PF-05251749: 10 mg + 100 mg + 500 mg + Placebo | Cohort 3 PF-05251749: 500 mg | Cohort 4 PF-05251749: 500 mg Unmilled + 500 mg Milled | Cohort 4 PF-05251749: 500 mg Milled + 500 mg Unmilled
Started | 1 | 2 | 2 | 3 | 2 | 2 | 2 | 2 | 0 | 0 | 0
Completed | 1 | 2 | 2 | 3 | 2 | 2 | 2 | 2 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Intervention Period 3 (3 Days)
Arm/Group | Cohort 1 PF-05251749: Placebo + 30 mg + 250 mg + 500 mg | Cohort 1 PF-05251749: 3 mg + Placebo + 250 mg + 500 mg | Cohort 1 PF-05251749: 3 mg + 30 mg + Placebo + 500 mg | Cohort 1 PF-05251749: 3 mg + 30 mg + 250 mg + Placebo | Cohort 2 PF-05251749: Placebo + 100 mg + 500 mg + 1000 mg | Cohort 2 PF-05251749: 10 mg + Placebo + 500 mg + 1000 mg | Cohort 2 PF-05251749: 10 mg + 100 mg + Placebo + 1000 mg | Cohort 2 PF-05251749: 10 mg + 100 mg + 500 mg + Placebo | Cohort 3 PF-05251749: 500 mg | Cohort 4 PF-05251749: 500 mg Unmilled + 500 mg Milled | Cohort 4 PF-05251749: 500 mg Milled + 500 mg Unmilled
Started | 1 | 2 | 2 | 3 | 2 | 2 | 2 | 2 | 0 | 0 | 0
Completed | 1 | 2 | 2 | 3 | 2 | 2 | 2 | 2 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 3 (7 Days)
Arm/Group | Cohort 1 PF-05251749: Placebo + 30 mg + 250 mg + 500 mg | Cohort 1 PF-05251749: 3 mg + Placebo + 250 mg + 500 mg | Cohort 1 PF-05251749: 3 mg + 30 mg + Placebo + 500 mg | Cohort 1 PF-05251749: 3 mg + 30 mg + 250 mg + Placebo | Cohort 2 PF-05251749: Placebo + 100 mg + 500 mg + 1000 mg | Cohort 2 PF-05251749: 10 mg + Placebo + 500 mg + 1000 mg | Cohort 2 PF-05251749: 10 mg + 100 mg + Placebo + 1000 mg | Cohort 2 PF-05251749: 10 mg + 100 mg + 500 mg + Placebo | Cohort 3 PF-05251749: 500 mg | Cohort 4 PF-05251749: 500 mg Unmilled + 500 mg Milled | Cohort 4 PF-05251749: 500 mg Milled + 500 mg Unmilled
Started | 1 | 2 | 2 | 3 | 2 | 2 | 2 | 2 | 0 | 0 | 0
Completed | 1 | 2 | 2 | 3 | 2 | 2 | 2 | 2 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Intervention Period 4 (3 Days)
Arm/Group | Cohort 1 PF-05251749: Placebo + 30 mg + 250 mg + 500 mg | Cohort 1 PF-05251749: 3 mg + Placebo + 250 mg + 500 mg | Cohort 1 PF-05251749: 3 mg + 30 mg + Placebo + 500 mg | Cohort 1 PF-05251749: 3 mg + 30 mg + 250 mg + Placebo | Cohort 2 PF-05251749: Placebo + 100 mg + 500 mg + 1000 mg | Cohort 2 PF-05251749: 10 mg + Placebo + 500 mg + 1000 mg | Cohort 2 PF-05251749: 10 mg + 100 mg + Placebo + 1000 mg | Cohort 2 PF-05251749: 10 mg + 100 mg + 500 mg + Placebo | Cohort 3 PF-05251749: 500 mg | Cohort 4 PF-05251749: 500 mg Unmilled + 500 mg Milled | Cohort 4 PF-05251749: 500 mg Milled + 500 mg Unmilled
Started | 1 | 2 | 2 | 3 | 2 | 2 | 2 | 2 | 0 | 0 | 0
Completed | 1 | 2 | 2 | 3 | 2 | 2 | 2 | 2 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population was defined as all participants who were randomized.
Groups:
- Cohort 1: Participants received a single oral dose of PF-05251749 suspension on Day 1 of each Intervention Period (4 Intervention Periods of 3 days each). Participants received study treatment in following sequences: Placebo, PF-05251749 30 mg, 250 mg and 500 mg; PF-05251749 3 mg, placebo, PF-05251749 250 mg and 500 mg; PF-05251749 3 mg, 30 mg, placebo and PF-05251749 500 mg; PF-05251749 3 mg, 30 mg, 250 mg and placebo in Intervention Period 1, 2, 3 and 4 respectively. All doses were administered in fasted state except PF-05251749 500 mg. A washout period of at least 7 days was maintained between each Intervention Period.
- Cohort 2: Participants received a single oral dose of PF-05251749 suspension on Day 1 of each Intervention Period (4 Intervention Periods of 3 days each). Participants received study treatment in following sequences: PF-05251749 placebo, PF-05251749 100mg, PF-05251749 500mg, PF-05251749 1000mg; PF-05251749 10mg, PF-05251749 placebo, PF-05251749 500mg, PF-05251749 1000mg; PF-05251749 10mg, PF-05251749 100mg, PF-05251749 placebo, PF-05251749 1000mg and PF-05251749 10mg, PF-05251749 100mg, PF-05251749 500mg, PF-05251749 placebo in Intervention Period 1, 2, 3 and 4 respectively. All doses were administered in fasted state. A washout period of at least 7 days was maintained between each Intervention Period.
- Cohort 3: Participants received a single oral dose of PF-05251749 500 mg suspension on Day 1. CSF samples were collected for a total of 10 hours beginning 2 hours predose and 8 hours post dose.
- Cohort 4: Participants received a single oral dose of PF-05251749 suspension on Day 1 of each Intervention Period (2 Intervention Periods of 3 days each). Participants received study treatment in following sequences: PF-05251749 500mg unmilled, PF-05251749 500mg milled and PF-05251749 500mg milled, PF-05251749 500mg unmilled in Intervention Period 1 and 2. All doses were administered in fasted state. A washout period of at least 7 days was maintained between each Intervention Period.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total
Number analyzed (Participants) | 9 | 11 | 6 | 6 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.7 (10.2) | 41.3 (6.3) | 44.5 (6.0) | 38.5 (11.2) | 38.9 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 9 | 11 | 6 | 6 | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: For Cohort 1 and 2: Baseline up to Week 8, Cohort 3: Baseline up to Week 2, Cohort 4: Baseline up to Week 3
Population: Safety analysis set included all participants who received at least 1 dose of study treatment.
Measure: Number; unit: participants
Groups:
- Cohort 1: PF-05251749 3 mg: Participants received a single oral dose of PF-05251749 3 mg oral suspension on Day 1 of Intervention Period in Cohort 1.
- Cohort 1: PF-05251749 30 mg: Participants received a single oral dose of PF-05251749 30 mg oral suspension on Day 1 of Intervention Period in Cohort 1.
- Cohort 1: PF-05251749 250 mg: Participants received a single oral dose of PF-05251749 250 mg oral suspension on Day 1 of Intervention Period in Cohort 1.
- Cohort 1: PF-05251749 500 mg (FED): Participants received a single oral dose of PF-05251749 500 mg oral suspension on Day 1 of Intervention Period in Cohort 1.
- Cohort 2: PF-05251749 10 mg: Participants received a single oral dose of PF-05251749 10 mg oral suspension on Day 1 of Intervention Period in Cohort 2.
- Cohort 2: PF-05251749 100 mg: Participants received a single oral dose of PF-05251749 100 mg oral suspension on Day 1 of Intervention Period in Cohort 2.
- Cohort 2: PF-05251749 500 mg: Participants received a single oral dose of PF-05251749 500 mg oral suspension on Day 1 of Intervention Period in Cohort 2.
- Cohort 2: PF-05251749 1000 mg: Participants received a single oral dose of PF-05251749 1000 mg oral suspension on Day 1 of Intervention Period in Cohort 2.
- Cohort 1-2: Placebo: Participants received a single oral dose of placebo matching to PF-05251749 oral suspension on Day 1 of Intervention Period in Cohort 1 and 2.
- Cohort 3: PF-05251749 500 mg CSF: Participants received a single oral suspension of PF-05251749 500 mg on Day 1. CSF samples were collected for a total of 10 hours beginning 2 hours predose and 8 hours post dose.
- Cohort 4: PF-05251749 500 mg Unmilled: Participants received a single oral dose of PF-05251749 10 mg oral suspension (unmilled) on Day 1 of Intervention Period in Cohort 4.
- Cohort 4: PF-05251749 500 mg Milled: Participants received a single oral dose of PF-05251749 10 mg oral suspension (milled) on Day 1 of Intervention Period in Cohort 4.
Arm/Group | Cohort 1: PF-05251749 3 mg | Cohort 1: PF-05251749 30 mg | Cohort 1: PF-05251749 250 mg | Cohort 1: PF-05251749 500 mg (FED) | Cohort 2: PF-05251749 10 mg | Cohort 2: PF-05251749 100 mg | Cohort 2: PF-05251749 500 mg | Cohort 2: PF-05251749 1000 mg | Cohort 1-2: Placebo | Cohort 3: PF-05251749 500 mg CSF | Cohort 4: PF-05251749 500 mg Unmilled | Cohort 4: PF-05251749 500 mg Milled
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15 | 6 | 6 | 6
participants | 0 | 2 | 0 | 1 | 0 | 0 | 4 | 3 | 3 | 5 | 0 | 1

2. Primary Outcome: Number of Participants With Laboratory Abnormalities
Description: Hemoglobin(Hgb),hematocrit,red blood cell(RBC):less than(<)0.8*lower limit of normal(LLN), MCV,MCH,MCHC,MPV:<0.9*LLN or >1.1*upper limit of normal(ULN), platelet:<0.5*LLN or >1.75*ULN, white blood cell(WBC):<0.6*LLNor>1.5*ULN, lymphocyte,neutrophil,total neutrophil:<0.8*LLN or >1.2*ULN,basophil,eosinophil,monocyte:>1.2*ULN; PTT, PT:>1.1*ULN,Fibrinogen<0.75*ULNor>1.25ULN; total, direct, indirect bilirubin >1.5*ULN,aspartate aminotransferase,alanine aminotransferase,gamma-glutamyl transferase,alkaline phosphatase:> 3.0*ULN,total protein,albumin:<0.8*LLN or >1.2*ULN;blood urea nitrogen,creatinine:>1.3*ULN,uric acid>1.2*ULN;sodium:<0.95*LLN or>1.05*ULN,potassium,chloride, calcium,magnesium,bicarbonate:<0.9*LLN or >1.1*ULN, phosphate<0.8*LLN or >1.2*ULN; glucose <0.6*LLN or >1.5*ULN,creatine kinase>2.0*ULN;urine(specific gravity<1.003or>1.030,pH <4.5or>8,glucose,ketone,protein,blood/Hgb,bilirubin,leukocyte esterase,crystals>=1,RBC,WBC >=20*ULN,bacteria>20);CSF (WBC>=6,RBC>0,Albumin>35).
Time Frame: Cohort 1 and 2: Baseline up to Week 8, Cohort 3: Baseline up to Week 2, Cohort 4: Baseline up to Week 3
Population: Safety analysis set included all participants who received at least 1 dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Cohort 1: PF-05251749 3 mg | Cohort 1: PF-05251749 30 mg | Cohort 1: PF-05251749 250 mg | Cohort 1: PF-05251749 500 mg (FED) | Cohort 2: PF-05251749 10 mg | Cohort 2: PF-05251749 100 mg | Cohort 2: PF-05251749 500 mg | Cohort 2: PF-05251749 1000 mg | Cohort 1-2: Placebo | Cohort 3: PF-05251749 500 mg CSF | Cohort 4: PF-05251749 500 mg Unmilled | Cohort 4: PF-05251749 500 mg Milled
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15 | 6 | 6 | 6
participants | 3 | 2 | 1 | 2 | 3 | 3 | 4 | 3 | 6 | 5 | 1 | 0

3. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Description: Criteria for clinically significant change from baseline in vital signs: supine systolic blood pressure (SBP) <90 millimeter of mercury (mmHg), supine diastolic BP (DBP) <50 mmHg, supine pulse rate <40 beats per minute (bpm) or >120 bpm. Maximum increase or decrease from baseline in supine SBP greater than or equal to (>=)30 mmHg and maximum increase or decrease from baseline in supine DBP >=20 mmHg.
Time Frame: Cohort 1 and 2: Baseline up to Week 8, Cohort 3: Baseline up to Week 2, Cohort 4: Baseline up to Week 3
Population: Safety analysis set included all participants who received at least 1 dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Cohort 1: PF-05251749 3 mg | Cohort 1: PF-05251749 30 mg | Cohort 1: PF-05251749 250 mg | Cohort 1: PF-05251749 500 mg (FED) | Cohort 2: PF-05251749 10 mg | Cohort 2: PF-05251749 100 mg | Cohort 2: PF-05251749 500 mg | Cohort 2: PF-05251749 1000 mg | Cohort 1-2: Placebo | Cohort 3: PF-05251749 500 mg CSF | Cohort 4: PF-05251749 500 mg Unmilled | Cohort 4: PF-05251749 500 mg Milled
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15 | 6 | 6 | 6
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Abnormal 12-Lead Electrocardiogram (ECG) Findings
Description: ECG parameters included maximum pulse rate (PR) interval, QRS interval, and corrected QT interval using Fridericia's formula (QTcF). Criteria for abnormal ECG: Maximum PR interval >=300 milliseconds (msec) or >=25 percent increase when baseline is >200 msec and >=50 percent increase when baseline is less than or equal to (=<) 200 msec; QRS interval >=140 msec or >=50 percent increase from baseline (IFB); and QTcF 30<=change<60 or change>=60 msec increase. The number of participants with abnormal ECG findings are reported.
Time Frame: Cohort 1 and 2: Baseline up to Week 8, Cohort 3: Baseline up to Week 2, Cohort 4: Baseline up to Week 3
Population: Safety analysis set included all participants who received at least 1 dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Cohort 1: PF-05251749 3 mg | Cohort 1: PF-05251749 30 mg | Cohort 1: PF-05251749 250 mg | Cohort 1: PF-05251749 500 mg (FED) | Cohort 2: PF-05251749 10 mg | Cohort 2: PF-05251749 100 mg | Cohort 2: PF-05251749 500 mg | Cohort 2: PF-05251749 1000 mg | Cohort 1-2: Placebo | Cohort 3: PF-05251749 500 mg CSF | Cohort 4: PF-05251749 500 mg Unmilled | Cohort 4: PF-05251749 500 mg Milled
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15 | 6 | 6 | 6
participants | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 2 | 1 | 0 | 0 | 1

5. Primary Outcome: Change From Baseline in Bond and Lader Visual Analogue Scale (BL-VAS) at 2 Hours Post Dose in Cohorts 1 and 2
Description: The BL-VAS monitored the subjective mood of each participant on 16 mood scales. Participants were asked to indicate on the VAS scale ranging from 0 to 100 mm about how they felt at the moment the scale was administered (example, alert/drowsy; calm/excited; content/tensed). The individual responses from the 16 mood scales were then combined to make three affective dimensions/subscales a) alertness (average of 9 items [total range 0 to 100, where each item is ordered so that higher scores indicated more alertness]), b) contentment (average of 2 items [total range 0 to 100, where higher scores indicated more contentment]), and c) calmness (average of 5 items [total range 0 to 100, where higher scores indicated more calmness]). Baseline is defined as the last available recording prior to dosing on Day 1 of the first Period.
Time Frame: Baseline, Day 1: 2 hours post dose
Population: Safety analysis set included all participants who received at least 1 dose of study treatment. This outcome measure was not planned to be analyzed in Cohort 3 and 4, as pre-specified in protocol.
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Cohort 1: PF-05251749 3 mg | Cohort 1: PF-05251749 30 mg | Cohort 1: PF-05251749 250 mg | Cohort 1: PF-05251749 500 mg (FED) | Cohort 2: PF-05251749 10 mg | Cohort 2: PF-05251749 100 mg | Cohort 2: PF-05251749 500 mg | Cohort 2: PF-05251749 1000 mg | Cohort 1-2: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15
millimeter
  Alertness: Baseline | 63.95 (21.656) | 83.05 (9.176) | 79.12 (21.139) | 74.92 (24.371) | 82.22 (14.773) | 89.98 (7.900) | 81.37 (22.535) | 87.57 (19.500) | 83.47 (14.945)
  Alertness: Change at 2 hours postdose | 11.48 (15.395) | 8.87 (20.227) | 8.65 (15.615) | 14.62 (23.859) | 2.28 (7.327) | 4.17 (3.247) | 0.30 (9.562) | -3.40 (10.744) | 7.45 (18.622)
  Calmness: Baseline | 68.83 (27.518) | 82.83 (10.424) | 84.67 (13.227) | 70.83 (23.962) | 73.58 (19.135) | 79.92 (21.280) | 90.33 (11.206) | 82.83 (19.372) | 80.10 (23.051)
  Calmness: Change at 2 hours postdose | 9.08 (14.857) | 12.42 (25.305) | 5.08 (5.800) | 2.33 (26.174) | 8.75 (6.594) | 5.42 (5.545) | 3.33 (7.878) | -10.33 (33.673) | 8.30 (25.787)
  Contentment: Baseline | 68.10 (26.737) | 83.20 (11.331) | 84.83 (11.542) | 78.03 (18.151) | 85.00 (14.105) | 84.63 (18.600) | 90.50 (9.294) | 89.70 (15.592) | 86.09 (16.013)
  Contentment: Change at 2 hours postdose | 7.57 (14.995) | 8.20 (21.017) | 5.20 (15.491) | 7.40 (29.055) | 4.90 (4.688) | 1.80 (5.362) | -0.43 (8.584) | -0.97 (11.598) | 5.55 (20.253)

6. Primary Outcome: Change From Baseline in Bond and Lader Visual Analogue Scale (BL-VAS) at 6 Hours Post Dose in Cohorts 1 and 2
Description: as for outcome 5
Time Frame: Baseline, Day 1: 6 hours post dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Cohort 1: PF-05251749 3 mg | Cohort 1: PF-05251749 30 mg | Cohort 1: PF-05251749 250 mg | Cohort 1: PF-05251749 500 mg (FED) | Cohort 2: PF-05251749 10 mg | Cohort 2: PF-05251749 100 mg | Cohort 2: PF-05251749 500 mg | Cohort 2: PF-05251749 1000 mg | Cohort 1-2: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15
millimeter
  Alertness: Change at 6 hours postdose | 9.25 (22.935) | 16.85 (16.053) | 12.72 (15.116) | 18.72 (22.991) | 3.43 (6.825) | -2.50 (18.228) | -1.07 (10.708) | -1.00 (8.820) | 5.93 (25.464)
  Calmness: Change at 6 hours postdose | 6.67 (7.916) | 6.83 (16.549) | -0.67 (16.136) | 16.00 (13.936) | 2.58 (6.829) | 8.33 (8.542) | -1.58 (16.209) | 2.17 (2.658) | 8.83 (25.441)
  Contentment: Change at 6 hours postdose | 7.53 (17.418) | 11.60 (19.555) | 4.80 (9.728) | 12.20 (23.074) | 1.20 (4.746) | 0.80 (9.955) | 0.40 (6.331) | 3.03 (9.063) | 7.51 (19.539)

7. Primary Outcome: Change From Baseline in Bond and Lader Visual Analogue Scale (BL-VAS) at 48 Hours Post Dose in Cohorts 1 and 2
Description: as for outcome 5
Time Frame: Baseline, Day 3: 48 hours post dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Cohort 1: PF-05251749 3 mg | Cohort 1: PF-05251749 30 mg | Cohort 1: PF-05251749 250 mg | Cohort 1: PF-05251749 500 mg (FED) | Cohort 2: PF-05251749 10 mg | Cohort 2: PF-05251749 100 mg | Cohort 2: PF-05251749 500 mg | Cohort 2: PF-05251749 1000 mg | Cohort 1-2: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15
millimeter
  Alertness: Change at 48 hours postdose | 15.83 (15.371) | 11.45 (13.703) | 15.80 (14.284) | 20.92 (19.343) | 3.90 (13.966) | 6.08 (7.372) | 6.12 (6.228) | 5.62 (6.576) | 9.67 (12.048)
  Calmness:Change at 48 hours postdose | -0.50 (23.791) | 6.17 (26.470) | 5.33 (9.983) | 8.67 (23.920) | 3.00 (5.550) | -4.83 (20.966) | -11.75 (25.284) | 10.00 (18.213) | 5.27 (18.547)
  Contentment: Change at 48 hours postdose | 13.70 (17.876) | 10.77 (16.112) | 6.87 (19.681) | 19.60 (21.045) | 4.00 (2.343) | 2.87 (3.090) | 4.60 (7.859) | 4.97 (5.967) | 7.56 (11.916)

8. Primary Outcome: Change From Baseline in Extrapyramidal Symptom Rating Scale (ESRS) at 2 Hours Post Dose in Cohorts 1 and 2
Description: ESRS is a clinician rated scale to assess parkinsonism,dystonia,dyskinesia,akathisia.The ESRS consists of 4 subscales and 4 clinicians global impressions-severity scales(CGI-S scales):I)a questionnaire of extrapyramidal symptoms or drug-induced movement disorders(a series of 4-point Likert scale questions with 0=Absent and 3=Severe);II)an examination of Parkinsonism and akathisia(7-point Likert scale with 0=Absent,6=extremely severe);III)an examination of dystonia(7-point Likert scale with 0=Absent,6=extremely severe);IV)an examination of dyskinesia(7-point Likert scale with 0=normal,6=most severe);V)toVIII)CGI-S scales(9-point Likert scale with 0=Absent,8=extremely severe)of tardive dyskinesia,parkinsonism,dystonia,akathisia.ESRS-Parkinsonism:total score range:0 to 14 where higher scores indicates greater severity;ESRS-dystonia:total score range:0 to 14 where higher scores indicates greater severity.Change from baseline was only observed in examination of parkinsonism and dystonia.
Time Frame: Baseline, Day 1: 2 hours post dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort 1: PF-05251749 3 mg | Cohort 1: PF-05251749 30 mg | Cohort 1: PF-05251749 250 mg | Cohort 1: PF-05251749 500 mg (FED) | Cohort 2: PF-05251749 10 mg | Cohort 2: PF-05251749 100 mg | Cohort 2: PF-05251749 500 mg | Cohort 2: PF-05251749 1000 mg | Cohort 1-2: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15
units on a scale
  Parkinsonism: Baseline | 0.0 (0.00) | 0.3 (0.52) | 0.3 (0.52) | 0.3 (0.52) | 0.2 (0.41) | 0.0 (0.00) | 0.2 (0.41) | 0.2 (0.41) | 0.1 (0.35)
  Parkinsonism: Change at 2 hours postdose | 0.0 (0.00) | 0.2 (0.75) | -0.3 (0.52) | -0.3 (0.52) | 0.2 (0.41) | 0.0 (0.00) | -0.2 (0.41) | -0.2 (0.41) | 0.0 (0.38)
  Dystonia: Baseline | 0.0 (0.00) | 0.2 (0.41) | 0.2 (0.41) | 0.2 (0.41) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.1 (0.26)
  Dystonia: Change at 2 hours postdose | 0.0 (0.00) | 0.0 (0.00) | -0.2 (0.41) | -0.2 (0.41) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)

9. Primary Outcome: Change From Baseline in Extrapyramidal Symptom Rating Scale (ESRS) at 48 Hours Post Dose in Cohorts 1 and 2
Description: as for outcome 8
Time Frame: Baseline, Day 1: 48 hours post dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort 1: PF-05251749 3 mg | Cohort 1: PF-05251749 30 mg | Cohort 1: PF-05251749 250 mg | Cohort 1: PF-05251749 500 mg (FED) | Cohort 2: PF-05251749 10 mg | Cohort 2: PF-05251749 100 mg | Cohort 2: PF-05251749 500 mg | Cohort 2: PF-05251749 1000 mg | Cohort 1-2: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15
units on a scale
  Parkinsonism:48 hours postdose | 0.0 (0.00) | 0.0 (0.63) | 0.0 (0.63) | -0.2 (0.41) | 0.2 (0.41) | 0.0 (0.00) | -0.2 (0.41) | -0.2 (0.41) | -0.1 (0.26)
  Dystonia: 48 hours postdose | 0.0 (0.00) | -0.2 (0.41) | -0.2 (0.41) | -0.2 (0.41) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)

10. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of PF-05251749
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours post dose
Population: The PK analysis set included all enrolled participants who were treated and had at least 1 measurable PK parameter of interest in at least 1 treatment period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Cohort 1: PF-05251749 3 mg | Cohort 1: PF-05251749 30 mg | Cohort 1: PF-05251749 250 mg | Cohort 1: PF-05251749 500 mg (FED) | Cohort 2: PF-05251749 10 mg | Cohort 2: PF-05251749 100 mg | Cohort 2: PF-05251749 500 mg | Cohort 2: PF-05251749 1000 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
nanogram per milliliter (ng/mL) | 16.7 (38) | 173.9 (33) | 1725 (39) | 1218 (33) | 60.08 (12) | 893.6 (32) | 3078 (18) | 4582 (35)
Statistical Analysis 1: Comparison: Cohort 1: PF-05251749 500 mg (FED) vs Cohort 2: PF-05251749 500 mg; Test type: Superiority or Other; Adjusted Geometric Mean Ratio. = 39.58, 90% CI 2-sided [30.14 to 51.99] — Values have been back-transformed from the log scale

11. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of PF-05251749
Description: Area under the plasma concentration-time profile from time zero to the time of last quantifiable concentration (Clast ).
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours post dose
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Cohort 1: PF-05251749 3 mg | Cohort 1: PF-05251749 30 mg | Cohort 1: PF-05251749 250 mg | Cohort 1: PF-05251749 500 mg (FED) | Cohort 2: PF-05251749 10 mg | Cohort 2: PF-05251749 100 mg | Cohort 2: PF-05251749 500 mg | Cohort 2: PF-05251749 1000 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
nanogram*hour per milliliter (ng*hr/mL) | 58.95 (52) | 714.7 (48) | 6542 (46) | 14120 (35) | 281.9 (19) | 3548 (27) | 17520 (23) | 33420 (36)
Statistical Analysis 1: Comparison: Cohort 1: PF-05251749 500 mg (FED) vs Cohort 2: PF-05251749 500 mg; Test type: Superiority or Other; Adjusted Geometric Mean Ratio = 80.60, 90% CI 2-sided [59.74 to 108.75] — Values have been back-transformed from the log scale

12. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] of PF-05251749
Description: AUC (0 -∞) = Area under the plasma concentration- time profile from time zero extrapolated to infinite time. It was calculated as AUC last + (C last*/k el), where C last* was the predicted plasma concentration at the last quantifiable time point estimated from the log-linear regression analysis.
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours post dose
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Cohort 1: PF-05251749 3 mg | Cohort 1: PF-05251749 30 mg | Cohort 1: PF-05251749 250 mg | Cohort 1: PF-05251749 500 mg (FED) | Cohort 2: PF-05251749 10 mg | Cohort 2: PF-05251749 100 mg | Cohort 2: PF-05251749 500 mg | Cohort 2: PF-05251749 1000 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
ng*hr/mL | 67.62 (50) | 729.2 (48) | 6607 (47) | 14350 (35) | 300.8 (19) | 3623 (27) | 17910 (24) | 33990 (36)
Statistical Analysis 1: Comparison: Cohort 1: PF-05251749 500 mg (FED) vs Cohort 2: PF-05251749 500 mg; Test type: Superiority or Other; Adjusted Geometric Mean Ratio = 80.12, 90% CI 2-sided [58.92 to 108.94] — Values have been back-transformed from the log scale

13. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-05251749
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours post dose
Population: The PK concentration analysis set included all enrolled participants who were treated and had at least 1 measurable concentration in at least 1 treatment period.
Measure: Median (Full Range); unit: hour
Arm/Group | Cohort 1: PF-05251749 3 mg | Cohort 1: PF-05251749 30 mg | Cohort 1: PF-05251749 250 mg | Cohort 1: PF-05251749 500 mg (FED) | Cohort 2: PF-05251749 10 mg | Cohort 2: PF-05251749 100 mg | Cohort 2: PF-05251749 500 mg | Cohort 2: PF-05251749 1000 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
hour | 1.00 [0.500 to 1.03] | 1.00 [0.500 to 1.50] | 1.00 [0.500 to 1.02] | 3.00 [0.500 to 8.00] | 1.00 [1.00 to 1.50] | 1.00 [0.500 to 1.00] | 1.25 [1.00 to 2.00] | 1.00 [1.00 to 4.00]

14. Secondary Outcome: Plasma Decay Half-Life (t1/2) of PF-05251749
Description: Terminal elimination half-life (t1/2). It was calculated as dividing the natural logarithm to the base e (Log e)*2/k el, where k el is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours post dose
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Cohort 1: PF-05251749 3 mg | Cohort 1: PF-05251749 30 mg | Cohort 1: PF-05251749 250 mg | Cohort 1: PF-05251749 500 mg (FED) | Cohort 2: PF-05251749 10 mg | Cohort 2: PF-05251749 100 mg | Cohort 2: PF-05251749 500 mg | Cohort 2: PF-05251749 1000 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
hour | 5.255 (2.5047) | 8.563 (3.3747) | 7.707 (2.3957) | 8.400 (1.1415) | 8.863 (2.2617) | 9.520 (2.6104) | 9.513 (2.1843) | 8.888 (1.2778)

15. Secondary Outcome: Apparent Oral Clearance (CL/F) of PF-05251749
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours post dose
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/hr)
Arm/Group | Cohort 1: PF-05251749 3 mg | Cohort 1: PF-05251749 30 mg | Cohort 1: PF-05251749 250 mg | Cohort 1: PF-05251749 500 mg (FED) | Cohort 2: PF-05251749 10 mg | Cohort 2: PF-05251749 100 mg | Cohort 2: PF-05251749 500 mg | Cohort 2: PF-05251749 1000 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
liter per hour (L/hr) | 44.38 (50) | 41.18 (48) | 37.87 (47) | 34.87 (35) | 33.25 (19) | 27.60 (27) | 27.90 (24) | 29.45 (36)

16. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of PF-05251749
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours post dose
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Cohort 1: PF-05251749 3 mg | Cohort 1: PF-05251749 30 mg | Cohort 1: PF-05251749 250 mg | Cohort 1: PF-05251749 500 mg (FED) | Cohort 2: PF-05251749 10 mg | Cohort 2: PF-05251749 100 mg | Cohort 2: PF-05251749 500 mg | Cohort 2: PF-05251749 1000 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Liter | 298.9 (37) | 458.5 (37) | 396.7 (29) | 419.0 (34) | 415.1 (22) | 365.7 (31) | 373.7 (18) | 374.4 (42)

17. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of Milled and Unmilled PF-05251749: Cohort 4
Description: Area under the plasma concentration-time profile from time zero to the time of last quantifiable concentration (Clast).
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours post dose
Population: The PK analysis set included all enrolled participants who were treated and had at least 1 measurable PK parameter of interest in at least 1 treatment period. This outcome measure was not planned to be analyzed for Cohort 1, 2 and 3, as pre-specified in protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Cohort 4: PF-05251749 500 mg Unmilled | Cohort 4: PF-05251749 500 mg Milled
Number analyzed (Participants) | 6 | 6
ng*hr/mL | 12600 (22) | 19210 (17)
Statistical Analysis 1: Comparison: Cohort 4: PF-05251749 500 mg Unmilled vs Cohort 4: PF-05251749 500 mg Milled; Test type: Superiority or Other; Adjusted Geometric Mean Ratio = 65.58, 90% CI 2-sided [62.18 to 69.16] — Values have been back-transformed from the log scale

18. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] of Milled and Unmilled PF-05251749: Cohort 4
Description: as for outcome 12
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours post dose
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Cohort 4: PF-05251749 500 mg Unmilled | Cohort 4: PF-05251749 500 mg Milled
Number analyzed (Participants) | 6 | 6
ng*hr/mL | 13440 (27) | 19590 (19)
Statistical Analysis 1: Comparison: Cohort 4: PF-05251749 500 mg Unmilled vs Cohort 4: PF-05251749 500 mg Milled; Test type: Superiority or Other; Adjusted Geometric Mean Ratio = 68.62, 90% CI 2-sided [63.27 to 74.41] — Values have been back-transformed from the log scale

19. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Milled and Unmilled PF-05251749: Cohort 4
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours post dose
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 4: PF-05251749 500 mg Unmilled | Cohort 4: PF-05251749 500 mg Milled
Number analyzed (Participants) | 6 | 6
ng/mL | 1007 (18) | 3385 (11)
Statistical Analysis 1: Comparison: Cohort 4: PF-05251749 500 mg Unmilled vs Cohort 4: PF-05251749 500 mg Milled; Test type: Superiority or Other; Adjusted Geometric Mean Ratio. = 29.76, 90% CI 2-sided [24.17 to 36.64] — Values have been back-transformed from the log scale

20. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Milled and Unmilled PF-05251749: Cohort 4
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours post dose
Population: as for outcome 17
Measure: Median (Full Range); unit: hour
Arm/Group | Cohort 4: PF-05251749 500 mg Unmilled | Cohort 4: PF-05251749 500 mg Milled
Number analyzed (Participants) | 6 | 6
hour | 2.50 [1.00 to 6.00] | 1.00 [0.500 to 1.00]

21. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Cerebrospinal Fluid (CSF) Concentration (AUClast) of PF-05251749
Description: Area under the CSF concentration-time profile from time zero to the time of last quantifiable concentration (Clast).
Time Frame: Predose, 1.5, 2.5, 4, and 8 hours post dose
Population: The PK analysis set included all enrolled participants who were treated and had at least 1 measurable PK parameter of interest in at least 1 treatment period. This outcome measure was not planned to be analyzed for Cohort 1, 2 and 4, as pre-specified in protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- Cohort 3: PF-05251749 500 mg (Plasma CSF Concentration): Participants received a single oral suspension of PF-05251749 500 mg on Day 1. CSF samples were collected for a total of 10 hours beginning 2 hours predose and 8 hours post dose.
- Cohort 3: PF-05251749 500 mg CSF: Participants received a single oral suspension of PF-05251749 500 mg on Day 1.
Arm/Group | Cohort 3: PF-05251749 500 mg (Plasma CSF Concentration) | Cohort 3: PF-05251749 500 mg CSF
Number analyzed (Participants) | 6 | 6
ng*hr/mL | 1824 (31) | 10920 (28)
Statistical Analysis 1: Comparison: Cohort 3: PF-05251749 500 mg (Plasma CSF Concentration) vs Cohort 3: PF-05251749 500 mg CSF; Test type: Superiority or Other; Adjusted Geometric Mean Ratio = 16.71, 90% CI 2-sided [15.35 to 18.18] — Values were back-transformed from the log scale

22. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Cerebrospinal Fluid (CSF) Infinite Time [AUC (0 - ∞)] of PF-05251749
Description: AUC (0 -∞) = Area under the CSF concentration- time profile from time zero extrapolated to infinite time. It was calculated as AUC last + (C last*/k el), where C last* was the predicted CSF concentration at the last quantifiable time point estimated from the log-linear regression analysis.
Time Frame: Predose, 1.5, 2.5, 4, and 8 hours post dose
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Cohort 3: PF-05251749 500 mg (Plasma CSF Concentration) | Cohort 3: PF-05251749 500 mg CSF
Number analyzed (Participants) | 6 | 6
ng*hr/mL | NA (NA) — Limited number of samples did not allow calculation of AUCinf; not analyzed. | NA (NA) — Limited number of samples did not allow calculation of AUCinf; not analyzed.

23. Secondary Outcome: Maximum Observed Cerebrospinal Fluid (CSF) Concentration (Cmax) of PF-05251749
Time Frame: Predose, 1.5, 2.5, 4, and 8 hours post dose
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 3: PF-05251749 500 mg (Plasma CSF Concentration) | Cohort 3: PF-05251749 500 mg CSF
Number analyzed (Participants) | 6 | 6
ng/mL | 354.6 (31) | 2331 (29)
Statistical Analysis 1: Comparison: Cohort 3: PF-05251749 500 mg (Plasma CSF Concentration) vs Cohort 3: PF-05251749 500 mg CSF; Test type: Superiority or Other; Adjusted Geometric Mean Ratio = 15.21, 90% CI 2-sided [13.29 to 17.42] — Values were back-transformed from the log scale

24. Secondary Outcome: Time to Reach Maximum Observed Cerebrospinal Fluid (CSF) Concentration (Tmax) of PF-05251749
Time Frame: Predose, 1.5, 2.5, 4, and 8 hours post dose
Population: as for outcome 21
Measure: Median (Full Range); unit: hour
Arm/Group | Cohort 3: PF-05251749 500 mg (Plasma CSF Concentration) | Cohort 3: PF-05251749 500 mg CSF
Number analyzed (Participants) | 6 | 6
hour | 1.59 [1.52 to 2.80] | 1.37 [1.37 to 4.00]

ADVERSE EVENTS:
Arm/Group | Cohort 1: PF-05251749 3 mg | Cohort 1: PF-05251749 30 mg | Cohort 1: PF-05251749 250 mg | Cohort 1: PF-05251749 500 mg (FED) | Cohort 2: PF-05251749 10 mg | Cohort 2: PF-05251749 100 mg | Cohort 2: PF-05251749 500 mg | Cohort 2: PF-05251749 1000 mg | Cohort 1-2: Placebo | Cohort 3: PF-05251749 500 mg CSF | Cohort 4: PF-05251749 500 mg Unmilled | Cohort 4: PF-05251749 500 mg Milled
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/15 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 2/6 | 0/6 | 1/6 | 0/6 | 0/6 | 4/6 | 3/6 | 3/15 | 5/6 | 0/6 | 1/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: PF-05251749 3 mg (N=6) | Cohort 1: PF-05251749 30 mg (N=6) | Cohort 1: PF-05251749 250 mg (N=6) | Cohort 1: PF-05251749 500 mg (FED) (N=6) | Cohort 2: PF-05251749 10 mg (N=6) | Cohort 2: PF-05251749 100 mg (N=6) | Cohort 2: PF-05251749 500 mg (N=6) | Cohort 2: PF-05251749 1000 mg (N=6) | Cohort 1-2: Placebo (N=15) | Cohort 3: PF-05251749 500 mg CSF (N=6) | Cohort 4: PF-05251749 500 mg Unmilled (N=6) | Cohort 4: PF-05251749 500 mg Milled (N=6)
Sinus node dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hunger (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vessel puncture site bruise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vessel puncture site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Procedural headache (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood pressure diastolic decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.